CLINICAL TRIAL: NCT00144105
Title: A Randomised, Open Label, Active Controlled Trial to Evaluate the Antiviral Efficacy and Safety of Treatment With 500 mg Tipranavir Plus 100 mg or 200 mg Ritonavir p.o. BID in Combination With Standard Background Regimen in Comparison to 400 mg Lopinavir Plus 100 mg Ritonavir p.o. BID in Combination With Standard Background Regimen in Antiretroviral Therapy Naive Patients for 48 With Extension up to 156 Weeks
Brief Title: A Randomised Trial to Evaluate the Antiviral Efficacy and Safety of Treatment With 500 mg Tipranavir (TPV) Plus 100 mg or 200 mg Ritonavir (RTV) p.o. BID in Comparison to 400 mg Lopinavir (LPV) Plus 100 mg RTV p.o. BID in Combination With Standard Background Regimen in ARV Therapy naïve Patients.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.33
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: TPV500mg/RTV200mgBID
Drug: TPV500mg/RTV100mgBID
Drug: LPV400mg/RTV100mgBID

SUMMARY:
Evaluation of safety and efficacy of Tipranavir (TPV) boosted with Ritonavir (RTV) versus an active control arm (Lopinavir / RTV) in antiretroviral (ARV) therapy naïve HIV-1 infected patients

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to trial participation.
2. HIV-1 infected males or females >= 18 years of age.
3. No previous ARV therapy.
4. Any CD4+ T lymphocyte count < 500 cells / µl.
5. HIV-1 viral load >= 5000 copies/mL at screening.
6. Screening laboratory values that indicate adequate baseline organ function.
7. A prior AIDS defining event is acceptable as long as it has resolved or the subject has been on stable treatment (e.g. opportunistic infection; no ARV) for at least 2 weeks before screening

Exclusion criteria:

1. Female patients of child-bearing potential who:

   * have a positive serum pregnancy test at screening or during the study,
   * are breast feeding,
   * are planning to become pregnant
2. Use of investigational medications within 30 days before study entry or during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2004-02; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of treatment responders at 48 weeks. A treatment responder is a patient with a viral load (VL) less than 50 copies/mL measured at two consecutive visits without prior rebound or change of ARV therapy.

SECONDARY OUTCOMES:
Further analyses to evaluate the primary endpoint at 24, 96, and 156 weeks. Secondary endpoints include proportion of patients with VL< 400 copies/mL, change from baseline in CD4+ cell counts at each visit, time to a new CDC class C progression event.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator
Locations (81):
- Argentina (4):
  - Boehringer Ingelheim Investigational Site, BsAs
  - Fundacion Huesped, Buenos Aires
  - Hospital de Agudos Teodoro Alvarez, Buenos Aires
  - Hospital Posadas, Haedo
- Australia (7):
  - Boehringer Ingelheim Investigational Site, Darlinghurst, New South Wales
  - St Vincents Hospital;, Darlinghurst, New South Wales
  - Boehringer Ingelheim Investigational Site, Liverpool, New South Wales
  - Boehringer Ingelheim Investigational Site, Surry Hills, New South Wales
  - Boehringer Ingelheim Investigational Site, Carlton, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Boehringer Ingelheim Investigational Site, South Yarra, Victoria
- Brazil (14):
  - Unidade de Pesquisa Clínica (UPC) - AIDS, Campinas - Sp
  - Boehringer Ingelheim Investigational Site, Curitiba - PR
  - Boehringer Ingelheim Investigational Site, Manguinhos - Rio de Janeiro - RJ
  - Instituto de Crianca / Hospital das Clínicas-FMUSP, Mooca / São Paulo
  - Hospital Geral de Nova Iguaçu - Ministério da Saúde, Nova Iguaçu - RJ
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro - RJ
  - Hospital Dia, Sacoma - São Paulo
  - Universidade Federal da Bahia-Unidade Docente Assistencial d, Salvador - BA
  - Boehringer Ingelheim Investigational Site, Santos - Sp
  - Hospital do Servidor Público Estadual de São Paulo, São Paulo - Sp
  - I.I. Emilio Ribas - Moléstias Infecciosas, São Paulo - SP
  - Instituto de Infectologia Emílio Ribas, São Paulo - SP
  - UNIFESP/ Hospital São Paulo- Univers. Federal de São Paulo, São Paulo - Sp
  - Centro de Referência e Treinamento - DST/AIDS, Vila Mariana - Sao Paulo
- Canada (12):
  - Downtown Infectious Diseases Clinic, Vancouver, British Columbia
  - Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - McMaster University Medical Centre, Hamilton, Ontario
  - The Ottawa Hospital Riverside Campus, Ottawa, Ontario
  - Canadian Immunodeficiency Research Collaborative Inc., Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook & Woman's College Health Science Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Whitby, Ontario
  - Montreal General Hospital - McGill University Health Centre, Monteal, Quebec
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Montreal Chest Institute, McGill University Health Centre, Montreal, Quebec
- Boehringer Ingelheim Investigational Site, Bogotá, Colombia
- France (7):
  - Hôpital Jean Verdier, Bondy
  - Hôpital Bocage, Dijon
  - Hôpital Albert Michallon, La Tronche
  - Hop Hôtel Dieu, Lyon
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Saint Antoine, Paris
  - Hôpital Bellevue, Saint-Etienne
- Germany (8):
  - Epimed GmbH, Berlin
  - Klinikum der Ruhr-Universität Bochum, Bochum
  - Universitätsklinik Köln, Cologne
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - ifi Studien und Projekte GbR, Hamburg
  - Medizinische Poliklinik, München
- Mexico (3):
  - Hospital de Especialidades no. 25, Col. Morelos, Monterrey, N. L.
  - Hospital Juan I. Menchaca IMSS, Col. Villaseñor, Guadalajara, Jal.
  - Hospital Lopez Mateos, México
- Poland (4):
  - Centre for AIDS Diagnostics and Therapy, Chorzów
  - Medical Academy of Szczecin, Szczecin
  - Hospital for Infectious Diseases, Warsaw
  - Department of Infectious Diseases, Wroclaw
- Romania (2):
  - Matei Bals Institute of Infectious Diseases, Bucharest
  - Victor Babes Clincial Hospital, Bucharest
- Russia (2):
  - Russian Federal Scientific, Moscow
  - City Hospital St Petersburg, Saint Petersburg
- Spain (11):
  - Boehringer Ingelheim Investigational Site, Badalona
  - Boehringer Ingelheim Investigational Site, Barcelona
  - Hospital Clínico y Provincial, Barcelona
  - Ciutat Sanitaria Universitaria de Bellvitge, Hospitalet de Llobregat (Barcelona)
  - Boehringer Ingelheim Investigational Site, Madrid
  - Hospital 12 de octubre, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Boehringer Ingelheim Investigational Site, Málaga
  - Boehringer Ingelheim Investigational Site, Santa Cruz de Tenerife
  - Hospital Universitario Vírgen del Rocío, Seville
  - Hospital Mútua de Terrasa, Terrassa
- Thailand (2):
  - Ramathibodhi Hospital, Bangkok
  - King Chulalonkorn Hospital, Pathumwan, Bangkok
- Princess Margaret Hospital, Nassau, The Bahamas
- United Kingdom (3):
  - Boehringer Ingelheim Investigational Site, Edinburgh
  - North Middlesex Hospital, London
  - Royal Free Hospital, London